CLINICAL TRIAL: NCT01048749
Title: Immediate Changes in Spinal Height and Pain Following Aquatic Vertical Suspension in Patients With Low Back Pain and Signs of Nerve Root Compression
Brief Title: Interventional Study of Effects on Spine Height With Two Unloading Positions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Jean Michel Brismee,PT, ScD Associate Professor, Texas Tech University Health Science Center
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: L08-144
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Low Back Pain
Keywords: Low back pain; nerve root compression; spinal height
MeSH Terms: conditions — Low Back Pain; Radiculopathy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aquatic vertical supsension (Active Comparator): Spinal height measurement using a stadiometer following aquatic vertical suspension
  Interventions: Other: aquatic vertical suspension.
- land-based supine flexion condition (Active Comparator): Spine height will be measured with a stadiometer following completion of the supine land-based flexion position.
  Interventions: Other: land-based supine flexion

INTERVENTIONS:
Other: aquatic vertical suspension. — Subject is suspended in a warm water deep pool with two pool noodles around the subject and directly under the axilla. Five pound weights are placed on the ankle and the subject maintains this unloaded position for 15 minutes.
  Other Names: Physical Therapy Treatment
  Arms: aquatic vertical supsension
Other: land-based supine flexion — The subject will lay supine with the legs supported by a foam wedge with hips flexed to 90 degrees and knees flexed to 65 degrees. They will maintain this unloaded position for 15 minutes.
  Other Names: Physical Therapy Treatment
  Arms: land-based supine flexion condition

SUMMARY:
The purpose of this study is to test a physical therapy intervention for reducing pain in the low back and into the legs. With individuals over the age of 40 years, this pain may be associated to changes in back height from aging of the cushions between the back bones. When pain is caused from this, completion of different positions and rest periods have been shown to help reduce the pain, at least temporarily. This study will compare two such positions; 1)floating in deep warm water with weights attached to the ankles, to take the load off of the spine, 2)lying on their back with hip and knees flexed to a 90 degree angle. The height of each person will be measured before and after completion of each intervention using a specially designed measuring tool.

Experimental hypothesis:

1. Subjects with low back and leg pain suggestive of nerve root compression syndrome will experience increase in spinal height when completing aquatic vertical suspension and/or land-based supine flexion.
2. Subjects with low back and leg pain suggestive of nerve root compression syndrome will experience greater increase in height, greater reduction of pain intensity and location when completing underwater vertical suspension as compared to supine land based flexion.

DETAILED DESCRIPTION:
Spinal height is affected throughout life from many different physiological changes and mechanical stresses, but a large portion is thought to occur primarily from intervertebral disc degeneration with resultant reduction in overall spinal height. The use of specific postures and rest periods to increase the overall spinal height has been suggested through various stadiometric research studies. This overall spinal height change can be used as a treatment tool for management of symptoms of chronic low back pain and signs of nerve root compression.

The purpose of the study is to investigate the effect of aquatic vertical suspension on spinal height, symptom location and pain intensity compared to a more commonly used land based supine flexion position.

The study will be conducted at one outpatient physical therapy clinic with subjects recruited from the local community.

A single blinded True Experimental Repeated Measure cross over design will be utilized.

Spine height will be measured using a commercially available stadiometer. Spinal height measurements will be completed after loaded walking, supine land based flexion positioning and after aquatic vertical hang.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 40-80 years,
* have current low back pain and/or numbness extending distal to the buttocks in the past 24 hours,
* pain level < 7/10 on the numerical rating scale, including symptom location change or pain intensity change with extension, lower limb weakness, achilles or patella reflex changes,
* reduction of lower limb sensation,
* positive SLR test.

Exclusion Criteria:

* inability to walk for a minimum of 15 minutes,
* inability to sit for a minimum of 5 minutes,
* inability to lie supine for a minimum of 15 minutes,
* fear of water or unwillingness to enter into a deep pool,
* allergy to chlorine,
* neurological disorders such as multiple sclerosis, spinal cord injury, incontinence, or spinal fusion,
* inability to elevate either shoulder above 90 degrees,
* pregnancy,
* vertebral fracture,
* pain level above 7/10 on the numeric pain scale or pain level reported at 0/10.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Differences of change of spinal height following aquatic vertical suspension compared to lumbar supine flexion positioning. | Spine height is measured prior to and after each intervention and then statistical comparisons completed.

SECONDARY OUTCOMES:
Differences in pain intensity and location following aquatic vertical suspension compared to supine land-based flexion position. | Pain intensity and location measurements are taken prior to and after completion of each intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jean M Brismee, PT, ScD, Study Chair — Texas Tech University Health Science Center; Susanne M Simmerman, PT, BS, Principal Investigator — Texas Tech University Health Science Center
Locations (1):
- Cleburne Physical Therapy and Fitness Center, Cleburne, Texas, United States